CLINICAL TRIAL: NCT02013557
Title: Text-message Reminders to Increase Rates of Postpartum Diabetes Screening in Women With Gestational Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources allocated elsewhere.
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Pro00015015
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes, Gestational
Keywords: Gestational Diabetes; Postpartum screening; Text-messages; 75-g oral glucose tolerance test
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Women in the intervention group will receive a test text-message reminder at the time of enrollment. They will then receive a text-reminder to schedule their oral glucose tolerance test at 6 weeks postpartum, with further reminders at 3 months and 6 months if they have not completed their testing.
  Interventions: Behavioral: Text-message reminder
- Control group (No Intervention): This arm will only receive the test text-message reminder at the time of enrollment. Otherwise they will receive usual postpartum care.

INTERVENTIONS:
Behavioral: Text-message reminder
  Arms: Intervention Group

SUMMARY:
Purpose: The purpose of this study is to see whether a text-message reminder system will increase the number of women who complete their diabetes screening after delivery.

Study Design: Prospective randomized control trial

Hypothesis: Gestational diabetics will be significantly more likely to follow up with their postpartum screening for diabetes if they receive text-message reminders to set up their lab appointment compared to those who receive usual care.

DETAILED DESCRIPTION:
Eligible participants will be recruited after delivery while on the postpartum ward. Recruitment will be conducted by the PI or a member of the study team. After informed consent is obtained, the patients will be randomized into one of two study groups: the intervention group or the control group. Women in the intervention group will receive a test text-message reminder at the time of enrollment. They will then receive a text-reminder to schedule their oral glucose tolerance test at 6 weeks postpartum, with further reminders at 3 months and 6 months if they have not completed their testing. Women in the control group will only receive the test text-message reminder. The PI or member of the study team obtaining the informed consent will verify the participant has received the text-message prior to completing enrollment. A computer-generated randomization list will be generated according to intervention vs. control group. Simple randomization will be used for the purposes of this study. 316 participants will be recruited based on the sample size calculations already performed. One group of 316 randomized opaque envelopes will be prepared. These sealed envelopes will be stored in a secured designated area at Tampa General Hospital. Once a patient has agreed to participate and is consented an envelope will be selected from the next sequentially numbered envelope and the number on the envelope will be recorded on their study sheet. Enrollment will continue until 316 participants have been recruited.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with gestational diabetes (GDM) based on a 100-g, 3-hour glucose tolerance test with 2 or more abnormal values according to the Carpenter-Coustan criteria OR Women with a 50-g, 1-hour loading test >200mg/dl.
* Diagnosed with GDM at least at 24 weeks gestation or later
* Access to a personal mobile phone with text-messaging capabilities.
* Age 18 or greater
* Able to provide written and informed consent in English or Spanish language

Exclusion Criteria:

* Women that were ever diagnosed with diabetes outside of pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that receive the 2-hour 75-g oral glucose tolerance test | Within six months of their delivery date

SECONDARY OUTCOMES:
Percentage of patients that receive any type of postpartum diabetes screening | Within six months of their delivery date
  This can include any of the multiple forms of diabetes screening tests including: 75-g oral glucose tolerance test, Hemoglobin A1c, fasting plasma glucose test or others.

CONTACTS AND LOCATIONS:
Overall Officials: Judette Louis, MD, Principal Investigator — University of South Florida Department of Obstetrics and Gynecology; Angela Gonzalez, MD, Study Chair — University of South Florida Department of Obstetrics and Gynecology
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No